CLINICAL TRIAL: NCT04273412
Title: Lifestyle Intervention for the Prevention of Gestational Diabetes Mellitus Among High-risk UAE Population
Brief Title: Lifestyle Intervention for Prevention of Gestational Diabetes Mellitus in the UAE Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rashid Centre for Diabetes and Research (Other)
Responsible Party: Principal Investigator, Dr.Amena Sadiya, Manager Dietetics, Rashid Centre for Diabetes and Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RCDR-GDM
Record Dates: First submitted 2020-02-09; First posted 2020-02-18 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lifestyle intervention (LI) (Experimental): moderate-intensity lifestyle intervention (Individualised counseling on diet, physical activity, and target weight gain) by license dietitian
  Interventions: Behavioral: moderate-intensity lifestyle intervention
- usual standard care group (UC) (No Intervention): standard antenatal care as per usual clinic protocol

INTERVENTIONS:
Behavioral: moderate-intensity lifestyle intervention — standardized 12- week program and would be delivered in 4 sessions (2 individual, 2 telephonic). This lifestyle modification program is a combination of diet therapy (optimum calorie), increased daily physical activity and behavioral modification (self-monitoring, stimulus control, motivational interviewing)
  Arms: lifestyle intervention (LI)

SUMMARY:
Gestational diabetes mellitus (GDM) is a high blood glucose (hyperglycemia) first occurring or first recognized during pregnancy, it is affecting 16.4% of women globally and 36.6 % in this region. It is consistent, strong evidence on the impact of GDM on short and long term health impacts on both mother and her child, thereby presenting significant challenges to acute care and public health. Currently, our understanding of strategies that are effective in preventing GDM is limited. Indeed, prospective studies have indicated a positive result of lifestyle intervention on preventing the risk of GDM in pregnant women but we lack consistency in the findings from randomized controlled trials (RCT). Moreover, most of these trials have been reported from developed countries and none of them were presented from this region. In the present project, we aim to determine whether GDM can be prevented by a 12-week moderate lifestyle intervention compared with usual standard care in high-risk pregnant women. In addition, we will also examine maternal pregnancy and birth outcomes.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is a high blood glucose (hyperglycemia) first occurring or first recognized during pregnancy, it is affecting 16.4% of women globally and 36.6 % in this region. It is consistent, strong evidence on the impact of GDM on short and long term health impacts on both mother and her child, thereby presenting significant challenges to acute care and public health. Currently, our understanding of strategies that are effective in preventing GDM is limited. Indeed, prospective studies have indicated a positive result of lifestyle intervention on preventing the risk of GDM in pregnant women but we lack consistency in the findings from randomized controlled trials (RCT). Moreover, most of these trials have been reported from developed countries and none of them were presented from this region. In the present project, we aim to determine whether GDM can be prevented by a 12-week moderate lifestyle intervention compared with usual standard care in high-risk pregnant women. In addition, we will also examine maternal pregnancy and birth outcomes. If the results show a positive association, we could develop this as a clinical process for improving patient care and cost.

This is a randomized controlled trial where participants will be included if they have more than one risk factors for GDM and randomized to two arms moderate-intensity lifestyle intervention (LI) or usual standard care group (control)(UC) between 6-12 gestational week. For the intervention group, standardized 12- week program and would be delivered in 4 sessions (2 individual, 2 telephonic) by a licensed dietitian. This lifestyle modification program is designed to achieve targeted weight gain and improve glycemic control through a combination of diet therapy, increased daily physical activity, and behavioral modification. The UC participants will receive no session as per the usual clinic protocol. Follow-up until l 24-28 gestational weeks, and the incidence of GDM was used to evaluate the effect of the intervention. At the end of interventions, participants in both arms will receive usual care based on their diagnosis and discretion of their physician. A sample size of 70 participants in each arm was estimated to give the power of 80%.

ELIGIBILITY:
Inclusion Criteria:

The study will include pregnant females (≤ 12 weeks of gestation), singleton pregnancy who meet ≥ 2 risk factors for GDM stated below:

* High Risk ethnic group (South Asian, Middle Eastern, Black Carribean)
* Family history of type 2 diabetes, especially in first-degree relatives
* previous macrosomic baby weighing >4.5 kg
* Body mass index greater than 30 kg/m2
* Previous history of GDM or polycystic ovarian syndrome

Exclusion Criteria:

* Any form of pregestational diabetes
* Fasting glucose > 126 mg/dL at first prenatal visit.
* Currently using corticosteroids, metformin or other medications interfering with glucose metabolism
* Psychiatric disorders
* Medical conditions preventing any physical exercise.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2018-10-13 (Actual); Primary Completion 2021-07-11 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
incidence of gestational diabetes mellitus | 24-28 weeks of gestation
  one or more pathological glucose values in a 75g, 2-h oral glucose tolerance test; fasting plasma glucose ≥ 5.3mmol/L, and 1-h value ≥ 8.6 mmol/L, and 2-h value ≥ 8.6 mmol/L

SECONDARY OUTCOMES:
feto-maternal outcomes | on delivery
  maternal weight gain
feto-maternall outcome | on delivery
  baby birth weight
feto-maternal | on delivery
  mode of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Amena Sadiya, Ph.D, Principal Investigator — Sheikh Khalifa Medical City Ajman
Locations (1):
- Rashid Centre for Diabetes and Research, Ajman, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sadiya A, Jakapure V, Shaar G, Adnan R, Tesfa Y. Lifestyle intervention in early pregnancy can prevent gestational diabetes in high-risk pregnant women in the UAE: a randomized controlled trial. BMC Pregnancy Childbirth. 2022 Aug 30;22(1):668. doi: 10.1186/s12884-022-04972-w. PMID 36042401